CLINICAL TRIAL: NCT06086639
Title: A PILOT TRIAL OF A FOUR SESSION ONLINE OCCUPATIONAL THERAPY GROUP TRANINIG FOR MOTHERS OF CHILDREN WITH FEEDING PROBLEMS
Brief Title: A FOUR SESSION ONLINE OCCUPATIONAL THERAPY GROUP TRANINIG FOR MOTHERS OF CHILDREN WITH FEEDING PROBLEMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Rukiye Begüm KOCA, Lecturer, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RKOCA
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Feeding and Eating Disorders; Child Behavior Problem; Feeding Behavior; Online Intervention; Occupational Therapy
Keywords: feeding and eating disorders; mother-child relations; online group intervention; occupational therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research group; mothers receiving online occupational therapy group training (Experimental): Participants in this group received online occupational therapy group training for 1 hour per week for 4 weeks.
  Session-1 Defining the problem Understanding the causes Oral motor structures and anomalies Discussion Session-2 Feedback sharing The relationship between feeding and sensory integration Recognizing the symptoms of sensory integration Disorders Strategies for sensory integration disorders Discussion Session-3 Feedback sharing Parent behaviors and attitudes Behavioral strategies for feeding problems Discussion Session-4 Feedback sharing Self-compassion and self-regulation Cope with stress Discussion Review of outputs
  Interventions: Other: Online Occupational Therapy Group Training
- Control group; Participants in this group did not receive any occupational therapy intervention duri (No Intervention): Participants in this group did not receive any occupational therapy intervention during the 4-week period.

INTERVENTIONS:
Other: Online Occupational Therapy Group Training — In this study, a 4-week online occupational therapy group training was conducted by an occupational therapist specialized in the field of nutrition. The content of the training, which takes place one hour a week, is given below; Session-1 Defining the problem Understanding the causes Oral motor structures and anomalies Discussion Session-2 Feedback sharing The relationship between feeding and sensory integration Recognizing the symptoms of sensory integration Disorders Strategies for sensory integration disorders Discussion Session-3 Feedback sharing Parent behaviors and attitudes Behavioral strategies for feeding problems Discussion Session-4 Feedback sharing Self-compassion and self-regulation Cope with stress Discussion Review of outputs
  Arms: Research group; mothers receiving online occupational therapy group training

SUMMARY:
Feeding problems such as selective eating, loss of appetite, and mealtime behavior problems are common in childhood. Parents play a primary role in learning about feeding, and difficulties experienced in this process may cause the parent to experience stress, despair and exhibit incorrect attitudes. The aim of this study is to examine the effect of online occupational therapy group training for mothers on mothers' attitudes and stress levels, and children's eating behaviors. Mothers of children aged 3-6 years with feeding problems (n=29) were randomly divided into groups. Early Childhood Adaptive Eating Behavior Scale, Feeding Process Mother Attitudes Scale and State-Trait Anxiety Inventory scales were used for evaluation. The mothers in the research group participated in the 4-week training. As a result of the research, positive effects were found on mothers' attitudes and children's eating behaviors (p<0.05). There was no change in mothers' state and trait anxiety levels (p>0.05). This study shows that online group training to mothers can support existing therapies and guides clinicians working in the field.

ELIGIBILITY:
Inclusion Criteria:

* Being a mother with a child between 37-72 months of age,
* Experiencing feeding problems with their child,
* Having the ability to understand the training and comprehend the scale items,
* Volunteering to participate,
* Having the competence to use online platforms, tools, and the internet connection.

Exclusion Criteria:

* Receiving special education and/or occupational therapy sessions due to any risk,
* Having any chronic disease or disability in their child.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female; Mothers with children between the ages of 3-6 can participate.
Enrollment: 29 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Early Childhood Adaptive Eating Behavior Scale | From enrollment to the end of treatment at 4 weeks
  Early Childhood Adaptive Eating Behavior Scale (ECAEBS), which was developed in 2018. The scale has a Cronbach's alpha value of 0.89, indicating good internal consistency, and a test-retest reliability coefficient of 0.96, indicating good stability over time. The scale consists of 20 items that are filled out by the caregiver and are rated on a 5-point Likert scale ranging from "Never" to "Always". The ECAEBS assesses various sub-factors, including "Reluctance," "Sensory-Related Rejection to Eat," "Aggression," and "Response to Main Meal Order." The total score of the scale can range from 20 to 100, with higher scores indicating a higher level of problems related to eating behaviors. An increase in scores for each sub-factor and the total score indicates an increase in feeding-related difficulties

SECONDARY OUTCOMES:
Feeding Process Mother Attitudes Scale | From enrollment to the end of treatment at 4 weeks
  Feeding Process Mother Attitudes Scale (FPMAS) to evaluate the attitudes of mothers in the process of feeding their children. This scale was developed in 2018 to assess mothers' feelings, thoughts, and approaches regarding the feeding process, specifically focusing on the interactional dimension of feeding with the mother. The FPMAS has a high internal consistency with a Cronbach's alpha value of 0.91 and good stability over time with a test-retest reliability coefficient of 0.94. The FPMAS is designed to evaluate the attitudes of mothers who have children between 9 months and 72 months old about the feeding process. It consists of 27 items rated on a 5-point Likert scale ranging from "Never" to "Always". The scale includes several sub-factors: "Negative Mood During Meal," "Attitudes towards Inadequate/Imbalanced Nutrition," "Negative Feeding Strategies," "Forced Feeding," and "Response to the Opinion of Others.". The total score on the FPMAS can range from 27 to 135

OTHER OUTCOMES:
State-Trait Anxiety Inventory | From enrollment to the end of treatment at 4 weeks
  State-Trait Anxiety Inventory (STAI), one of the most widely used scales in the health field, to assess the anxiety level of mothers. The STAI consists of two separate scales, each consisting of forty items, making a total of eighty items. The State Anxiety Inventory measures how the person feels at a certain moment, reflecting their current state of anxiety. On the other hand, the Trait Anxiety Inventory measures how the person generally feels, providing an insight into their overall trait anxiety. Both scales can be completed in a total of 20 minutes. The interpretation of scores is done based on the total score obtained from both inventories, which can range between 20 and 80. A high score indicates a high level of anxiety, while a low score indicates a low level of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Ankara/ Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Concern that there is a risk of losing control of the data and that the data may be misused and unfair benefit may be obtained from the data.